CLINICAL TRIAL: NCT01841229
Title: Effect of Ginseng on Glycemic Control: A Systematic Review and Meta-analysis of Controlled Trials to Provide Evidence-based Clinical Recommendations
Brief Title: Effect of Ginseng on Glycemic Control
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: MetaG
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Impaired Glucose Tolerance; Diabetes
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Ginseng (American ginseng, Asian ginseng, Korean ginseng etc) is expected to show positive hypoglycemic effects, including improvements in glycated blood proteins[HbA1c], fasting glucose, fasting insulin, and the homeostasis model assessment of insulin resistance [HOMA-IR]).

DETAILED DESCRIPTION:
Ginseng has demonstrated to have significant hypoglycemic effect. Its major pharmacological component is considered to be ginsenosides. Several trials have been undertaken in diabetes some of which have demonstrated advantages in glycemic control in both diabetic as well as non diabetic individuals although clinical consistency of results is lacking.The lack of high quality data in this area to support diabetes recommendations represents an urgent call for stronger evidence. A systematic review and meta-analysis of controlled trials remains the "Gold Standard" of evidence for recommendations and clinical guidelines development. Therefore, investigators will conduct a systematic review and meta-analyses of controlled trials to assess the effect of ginseng on glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized treatment allocation
* 1 month
* Suitable control
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* Non-randomized treatment allocation
* <1 month
* Lack of a suitable control
* No viable endpoint data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Diabetic (type 1 & type 2) Pre-diabetic Hypertensive Healthy
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 1month

SECONDARY OUTCOMES:
Fasting blood glucose | 1month
Fasting plasma insulin | 1 month
Homeostasis model assessment of insulin resistance (HOMA-IR) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St.Michael's Hospital., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Shishtar E, Sievenpiper JL, Djedovic V, Cozma AI, Ha V, Jayalath VH, Jenkins DJ, Meija SB, de Souza RJ, Jovanovski E, Vuksan V. The effect of ginseng (the genus panax) on glycemic control: a systematic review and meta-analysis of randomized controlled clinical trials. PLoS One. 2014 Sep 29;9(9):e107391. doi: 10.1371/journal.pone.0107391. eCollection 2014. PMID 25265315